CLINICAL TRIAL: NCT06699784
Title: Quality of Life in Presbyopes Using Single-vision Lens and Progressive Lens Correction: a Randomized Controlled Trial
Brief Title: Quality of Life in Presbyopes Using Single-vision Lens and Progressive Lens Correction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20240916011
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Presbyopia; Presbyopia Correction
Keywords: quality of life; presbyopia; near correction
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Progressive lenses intervention group (Experimental): Progressive lenses intervention group will receive 1-month progressive lens correction in daily life.
  Interventions: Behavioral: Progressive lenses intervention
- Single-vision lenses intervention group (Placebo Comparator): Single-vision lenses intervention group will use near-vision spectacles during near work and use their original habitual distant glasses for distance tasks for 1 month.
  Interventions: Behavioral: Single-vision lenses intervention

INTERVENTIONS:
Behavioral: Progressive lenses intervention — Progressive lenses intervention group will receive 1-month progressive lens correction in daily life.
  Arms: Progressive lenses intervention group
Behavioral: Single-vision lenses intervention — Single-vision lenses intervention group will use near-vision spectacles during near work and use their original habitual distant glasses for distance tasks for 1 month.
  Arms: Single-vision lenses intervention group

SUMMARY:
The goal of this clinical trial is to compare the quality of life (QOL) of presbyopes wearing progressive addition lenses (PALs) with that of those wearing single-vision spectacles (SVSs) for near correction. The main questions it aims to answer is:

What is the difference in QOL between presbyopes who use SVSs and those who use PALs ? Eligible participants will be randomly assigned in a 1:1 ratio to either the PALs group or the SVSs group.Participants in the progressive lenses intervention group will receive 1-month progressive lens correction in daily life. And participants in single-vision lenses intervention group will use near-vision spectacles during near work and use their original habitual distant glasses for distance tasks for 1 month.

The study will compare the QOL scores measured by a 12-item Near Vision-Related Quality of Life questionnaire between the two groups. Additionally, the study will compare the scores measured by the Refractive Status and Vision Profile questionnaire and Visual Analogue Scale questionnaire between the two groups as well as assess the change in the above three questionnaires scores at 1 month following enrollment. And visual acuity of subjects will also be assessed at baseline and at the 1-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40-70 years;
2. A distant correction of ≤2D for hyperopia, or >-2 D for myopia, or < 2D for astigmatism in both eyes;
3. Anisometropia of less than 1.50 D;
4. Distance best-corrected visual acuity (BCVA) of at least 0.5 LogMAR, and near VA < N8 (20/50) at 40 cm with habitually worn distance refractive correction, with improvement of near vision by at least one line on a near LogMAR E chart with the use of a plus lens;
5. Have not undergone any near correction in the past six months;
6. Able to answer a questionnaire;
7. Giving written consent to participate in the study.

Exclusion Criteria:

1. Ocular abnormalities leading to visual impairment including severe cataract, glaucoma, strabismus, and ocular fundus diseases;
2. Severe physiological and psychological diseases affecting follow-up;
3. History of cataract surgery, phakic intraocular lens surgery, corneal surgery, or any intraocular surgery affecting the refractive status of the eye;
4. Have used pilocarpine in the past six months.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
quality of life score | From enrollment to the end of intervention at 1 month
  Quality of life scores measured by a 12-item Near Vision-Related Quality of Life questionnaire.

SECONDARY OUTCOMES:
Other questionnaire | From enrollment to the end of intervention at 1 month
  •The scores of the refractive status and vision profile (RSVP) questionnaire and visual analogue scale (VAS).
Visual acuity | From enrollment to the end of intervention at 1 month
  Near and distance best-corrected visual acuity.

IPD SHARING:
Plan to Share IPD: No